CLINICAL TRIAL: NCT07063342
Title: Phase 1, 3-Part, Open-label Study to Evaluate the Pharmacokinetics of Novel KarX (BMS-986519) and KarT (BMS-986520) Prototypes Versus the KarXT (BMS-986510) and KarX-EC (BMS-986519) Reference Following Single Doses, and to Explore the Effect of Food After Multiple Doses of Selected Prototypes in Healthy Adult Participants
Brief Title: A Study to Evaluate Novel KarX and KarT Prototypes Versus the KarXT and KarX-EC Reference Following Single Doses, and to Explore the Effect of Food After Multiple Doses of Selected Prototypes in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0043; U1111-1321-3511 (Other: WHO)
Record Dates: First submitted 2025-06-23; First posted 2025-07-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride Capsule; Drug: Xanomeline Enteric Capsule; Drug: Trospium Chloride
- Part 2 (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride Capsule; Drug: Xanomeline Enteric Capsule; Drug: Trospium Chloride
- Part 3 (Experimental)
  Interventions: Drug: Xanomeline/Trospium Chloride Capsule; Drug: Xanomeline Enteric Capsule

INTERVENTIONS:
Drug: Xanomeline/Trospium Chloride Capsule — Specified dose on specified days
  Other Names: BMS-986510; KarXT
Drug: Xanomeline Enteric Capsule — Specified dose on specified days
  Other Names: BMS-986519; KarX-EC
Drug: Trospium Chloride — Specified dose on specified days
  Other Names: BMS-986520; KarT
  Arms: Part 1; Part 2

SUMMARY:
The purpose of this study is to evaluate novel KarX and KarT prototypes versus the KarXT and KarX-EC reference following single doses, and to explore the effect of food after multiple doses of selected prototypes in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 kg/m2 to 32.0 kg/m2, inclusive, at screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 23
Time of maximum observed concentration (Tmax) | Up to Day 23
Area under the concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to Day 23
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | Up to Day 23
Area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to Day 23
Concentration at the end of a dosing interval (Ctau) | Up to Day 23
Apparent total body clearance (CLT/F) | Up to Day 23
Effective elimination half-life during dosing interval (T-HALF(eff)) | Up to Day 23

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | Up to 30 days after final dose of study intervention
Number of participants with Serious Adverse Events (SAEs) | Up to 30 days after final dose of study intervention
Number of participants with Adverse Events of Special Interest (AESIs) | Up to 30 days after final dose of study intervention
Number of participants with AEs leading to discontinuation | Up to 30 days after final dose of study intervention
Number of participants with vital signs abnormalities | Up to 30 days after final dose of study intervention
Number of participants with electrocardiogram (ECG) abnormalities | Up to 30 days after final dose of study intervention
Number of participants with physical examination abnormalities | Up to 30 days after final dose of study intervention
Number of participants with clinical laboratory abnormalities | Up to 30 days after final dose of study intervention
Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to Day 25
Geometric mean ratio of Cmax | Up to Day 23
Geometric mean ratio of AUC(0-T) | Up to Day 23
Geometric mean ratio of AUC(INF) | Up to Day 23
Geometric mean ratio of area under the concentration-time curve in 1 dosing interval (AUC(TAU)) | Up to Day 23

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Quotient Sciences, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html